CLINICAL TRIAL: NCT06710717
Title: Autologous CD19 Car T-Cell Therapy For Patients With Severe Refractory Systemic Lupus Erythematosus - A Pilot Study
Brief Title: Autologous CD19 Car T-Cell Therapy For Severe Refractory Systemic Lupus Erythematosus (SLE)
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: National University of Malaysia (Other)
Collaborators: Plutonet Sdn Bhd (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: JEP-2024-754
Record Dates: First submitted 2024-11-21; First posted 2024-11-29 (Actual); Last update posted 2025-05-29 (Actual); Status verified 2025-05

CONDITIONS: Systemic Lupus Erythematous (SLE)
Keywords: CAR T cells; SLE; treatment-refractory; severe SLE
MeSH Terms: conditions — Lupus Erythematosus, Systemic

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- autologous CD19 CAR T-cells (Experimental): Single Infusion of autologous CD19 CAR T- cells
  Interventions: Biological: CD19 CAR-T cells

INTERVENTIONS:
Biological: CD19 CAR-T cells — Study participant will be given single infusion of autologous CD19 CAR-T cells following lymphodepletion chemotherapy

SUMMARY:
This pilot clinical study aims to evaluate the effectiveness of Chimeric Antigen Receptor (CAR) T-cell therapy in treating severe, refractory systemic lupus erythematosus (SLE), an autoimmune disease driven by autoreactive B-cells. Current treatments for severe SLE, including glucocorticoids, cytotoxic, and immunosuppressive drugs, have significant limitations. These treatments do not adequately control the underlying autoimmune process and require long-term use, leading to chronic side effects and often failing to prevent permanent organ damage. Given the high prevalence and mortality rates associated with SLE in regions like Asia and Malaysia, there is a pressing need for more effective therapies.

DETAILED DESCRIPTION:
This study seeks to investigate CAR-T cell therapy's potential for treating severe treatment-refractory systemic lupus erythematosus (SLE) in Malaysian patients.

STUDY OBJECTIVES

General Objective: To evaluate the safety and efficacy of autologous CD19 CAR T-cell infusion in patients with severe refractory SLE.

Specific Objectives:

To evaluate the safety and tolerability of treatment. To evaluate efficacy as measured by response rates and survival. To evaluate the quality of life based on the use of validated health questionnaire tools.

Hypothesis:

Intravenous autologous CD19 CAR T-cell therapy is safe, and efficacious in patients with severe refractory SLE.

EXPECTED OUTCOME OF THE STUDY:

CD19 CAR T-cell therapy is expected to result in:

Clinical remission as assessed by DORIS remission) with a good safety profile Serologic remission (defined as negative anti-dsDNA and normal complement C3 and C4 levels) at 3 months Sustained DORIS remission for at least 12 months Improvement in organ function Prolongation of duration of drug-free remission Improvement in quality of life Manageable adverse effects

STUDY POPULATION This pilot study will be conducted between 2025 and 2028 involving 5 patients diagnosed with severe, treatment-refractory SLE. Eligibility criteria were based on previously published studies and international guidelines for CAR treatment for patients with autoimmune disease (Boulougoura et al., 2023).

ELIGIBILITY:
Inclusion Criteria:

-

Aged between ≥ 18 to ≤ 65 years Clinical Diagnosis of SLE according to the 2019 European League Against Rheumatism/American College of Rheumatology (EULAR/ACR) classification criteria (Fanouriakis et al., 2019) Positive anti-nuclear antibody (ANA) (titer ≥1:80 ), anti-dsDNA (≥30 IU/mL on enzyme-linked immunosorbent assay [ELISA]), or anti-Smith at screening or by documented medical history Active disease (defined by not being in remission according to DORIS criteria or in a low disease activity state [LLDAS]) (Franklyn et al., 2016, van Vollenhoven et al., 2021) With at least one active organ system involvement Persistent active disease with insufficient response to glucocorticoids and at least 2 of the following treatments for at least 3 months each: cyclophosphamide, mycophenolate mofetil or its derivatives, belimumab, azathioprine, anifrolumab, methotrexate, rituximab, obinutuzumab, cyclosporin, tacrolimus or voclosporin.

Serum ALT <5 times the normal value, serum bilirubin <3 times the normal value, Left ventricular ejection fraction >45% Life expectancy of more than 3 months Eastern Cooperative Oncology Group (ECOG) performance status ≤2. Psychological, sociological or geographical conditions precluding compliance A female of childbearing age must have a negative pregnancy test and is on two effective contraception methods A male must use two effective contraception methods

Exclusion Criteria:

-

Active cancer or receiving cancer treatment Evidence of severe lung, FVC <45% and/or DLCO (corrected for Hb) <30% predicted, heart (NYHA class III/IV, arrhythmia, AV block, uncontrolled hypertension), liver failure or severe neurologic disorders.

Pre-existing irreversible kidney damage and creatinine clearance below 30 ml/min ( to review) Severe pancytopenia HIV positivity. Active Hepatitis B, C infection. Septicemia. Pregnant/nursing female. Receiving stem cell transplant within 12 weeks of enrolment, chemotherapy or radiotherapy within 8 weeks of enrolment Active CNS involvement.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Estimated)
Dates: Start 2025-01-03 (Actual); Primary Completion 2028-12-02 (Estimated); Study Completion 2029-01-02 (Estimated)

PRIMARY OUTCOMES:
Rate of Adverse events | Starting form day 0 up to 24 months after CAR-T cells infusion
  Incidence of adverse event (AE), classified according to CTCAE version 5.0, and evaluation and classification of Cytokine Release Syndrome (CRS) and Immune Effector cell-associated Neurotoxicity Syndrome (ICANS)
SLEDAI Remission Rate | Weeks 4, 8, 12, 16, 20, 24,28 after CAR-T cells infusion
  Remission is evaluated by fulfilment of SLEDAI remission criteria

SECONDARY OUTCOMES:
Clinical Response Rate | Weeks 4, 8, 12, 16, 20, 24,28 after CAR-T cells infusion
  Measured by BILAG, PGA, SLICC/ACR
Rate of B cell aplasia | Months 1, 3, 6, 9, 12, 15, 18, 21, 24 after CAR-T cells infusion
  Numbers of B cells in peripheral blood measured by flow cytometry
Rate of Immunological response | Months 1, 3, 6, 9, 12, 15, 18, 21, 24 after CAR-T cells infusion
  Changes in the levels of SLE-associated serum autoantibodies
Mean of Quality of life score | Weeks 4, 8, 12, 16, 20, 24,28 after CAR-T cells infusion
  Quality of life Assessed by FACIT-F

CONTACTS AND LOCATIONS:
Locations (1):
- University Kebangsaan Malaysia Medical Center, Bandar Tun Razak, Kuala Lumpur, Malaysia

IPD SHARING:
Plan to Share IPD: No